CLINICAL TRIAL: NCT03922659
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation and Cognitive Behavioral Therapy on Heroin Dependence
Acronym: THED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Peng, Professor, Director of Department of Neurology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-12-TMSCBT-H
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Heroin Dependence
Keywords: Heroin dependence, transcranial magnetic stimulation, cognitive behavioral therapy
MeSH Terms: conditions — Heroin Dependence | interventions — Transcranial Magnetic Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Regular treatment (symptomatic treatment) with blank TMS (Placebo Comparator): Regular treatment (symptomatic treatment) with blank transcranial magnetic stimulation
  Interventions: Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy
- Regular treatment (RT) with blank TMS and CBT (Active Comparator): Regular treatment (symptomatic treatment) with blank transcranial magnetic stimulation and cognitive behavioral therapy
  Interventions: Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy
- RT with right DLPFC hf-rTMS (Active Comparator): Regular treatment with right dorsolateral prefrontal cortex (DLPFC) high frequency repetitive transcranial magnetic stimulation (hf-rTMS)
  Interventions: Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy
- RT with right DLPFC hf-rTMS and CBT (Active Comparator): Regular treatment with right DLPFC high frequency repetitive transcranial magnetic stimulation (hf-rTMS) and cognitive behavioral therapy (CBT)
  Interventions: Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy
- RT with left DLPFC hf-rTMS (Active Comparator): Regular treatment with left DLPFC high frequency repetitive transcranial magnetic stimulation (hf-rTMS)
  Interventions: Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy
- RT with left DLPFC hf-rTMS and CBT (Active Comparator): Regular treatment with left DLPFC high frequency repetitive transcranial magnetic stimulation (hf-rTMS) and cognitive behavioral therapy (CBT)
  Interventions: Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy

INTERVENTIONS:
Combination Product: Transcranial magnetic stimulation and Cognitive behavioral therapy — Transcranial magnetic stimulation on different side with/without cognitive behavioral therapy

SUMMARY:
Heroin dependence is one of most common substance dependence, which brings great burden on health worldwide. Heroin dependence may lead to immunosuppression and cognitive impairments. Once heroin dependence is developed, it will be difficult to recover and easy to relapse. Although many efforts had been made in the treatment of heroin dependence, the annual recurrence of heroin dependence with traditional therapies would be up to 90%. Repetitive transcranial magnetic stimulation (rTMS) on the dorsolateral prefrontal cortex (DLPFC) or cognitive behavioral therapy (CBT) each alone was reported to have some effect on preventing from relapse of substance dependence. In order to test whether combined therapy of high frequency rTMS (hf-rTMS) with CBT is better for preventing from relapse of heroin dependence, we recruit patients with heroin dependence to participate this study. The study is a factorial designed and the patients will be assigned into one of the following six groups randomly: (1) regular treatment (symptomatic treatment) with blank TMS; (2) regular treatment (RT) with blank TMS and CBT; (3) RT with right DLPFC hf-rTMS; (4) RT with right DLPFC hf-rTMS and CBT; (5) RT with left DLPFC hf-rTMS; (6) RT with left DLPFC hf-rTMS and CBT. TMS was given 5 days per week for total 2 weeks using uniform scheme (5 seconds of 10Hz stimulation per train, 30 trains per day with inter-train interval of 20 seconds). CBT will be given once per week for total 8 weeks. The patients will be followed up for 6 months. Recurrence of heroin dependence, duration of abstention, heroin/drug intake, craving for heroin and other cognitive psychological assessments will be recorded and compared among the 6 treatment groups and the efficacy of combined therapy of rTMS with CBT will be evaluated in our study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as heroin dependence according to DSM-IV criteria
* No definite history of neurological diseases and psychological problems
* Volunteer to participate the study, cooperate to be followed up

Exclusion Criteria:

* Acute withdrawal state and CIWA score > 9
* With other neurological diseases and psychological problems
* With ever brain trauma and damage
* With other psychological medications or other substance dependence
* With other contraindications to have transcranial magnetic stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of heroin dependence | 1 month
  The rate of relapse of heroin dependence after discharge from hospital
Recurrence of heroin dependence | 2 month
  The rate of relapse of heroin dependence after discharge from hospital
Recurrence of heroin dependence | 3 month
  The rate of relapse of heroin dependence after discharge from hospital
Recurrence of heroin dependence | 6 month
  The rate of relapse of heroin dependence after discharge from hospital

SECONDARY OUTCOMES:
Duration of abstinence | 6 months
  The total time or period without any intake of heroin during follow-ups
Heroin consumption | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Diaries of heroin intake in different time of the follow-ups
Craving for heroin | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Craving assessment for heroin by Heroin Craving Questionnaire (HCQ) ranging from 0 to 175. Higher score of HCQ indicates more desire for heroin.
Craving for heroin | 2weeks, 1 month, 2 months, 3 months and 6 months
  Craving assessment by Visual Analogue Scale (VAS) for heroin desire ranging 0 to 10. Higher score indicates more desire for heroin.
Cognitive assessment | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Cognitive assessment by Montreal Cognitive Assessment (MoCA) ranging from 0 to 30. Lower score indicates worse cognitive function.
Psychological assessment - Anxiety | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Psychological assessment by Generalized Anxiety Disorder-7 (GAD-7) ranging from 0 to 21. Higher score indicates more severer anxiety.
Psychological assessment - Depression | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Psychological assessment by Patient Health Questionnaire-9 (PHQ-9) ranging from 0 to 27. Higher score indicates more severer depression.
Psychological assessment - Sleep | 2 weeks, 1 month, 2 months, 3 months and 6 months
  Psychological assessment by Pittsburgh Sleep Quality Index (PSQI) ranging from 0 to 21. Higher score indicates worse sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips MR, Zhang J, Shi Q, Song Z, Ding Z, Pang S, Li X, Zhang Y, Wang Z. Prevalence, treatment, and associated disability of mental disorders in four provinces in China during 2001-05: an epidemiological survey. Lancet. 2009 Jun 13;373(9680):2041-53. doi: 10.1016/S0140-6736(09)60660-7. PMID 19524780
- [Background] Makani R, Pradhan B, Shah U, Parikh T. Role of Repetitive Transcranial Magnetic Stimulation (rTMS) in Treatment of Addiction and Related Disorders: A Systematic Review. Curr Drug Abuse Rev. 2017;10(1):31-43. doi: 10.2174/1874473710666171129225914. PMID 29189190
- [Background] Shen Y, Cao X, Tan T, Shan C, Wang Y, Pan J, He H, Yuan TF. 10-Hz Repetitive Transcranial Magnetic Stimulation of the Left Dorsolateral Prefrontal Cortex Reduces Heroin Cue Craving in Long-Term Addicts. Biol Psychiatry. 2016 Aug 1;80(3):e13-4. doi: 10.1016/j.biopsych.2016.02.006. Epub 2016 Feb 12. No abstract available. PMID 26995024
- [Background] Herremans SC, Vanderhasselt MA, De Raedt R, Baeken C. Reduced intra-individual reaction time variability during a Go-NoGo task in detoxified alcohol-dependent patients after one right-sided dorsolateral prefrontal HF-rTMS session. Alcohol Alcohol. 2013 Sep-Oct;48(5):552-7. doi: 10.1093/alcalc/agt054. Epub 2013 May 24. PMID 23709633